CLINICAL TRIAL: NCT01397643
Title: A Prospective Randomised Trial of Non-operative Versus Operative Management of Olecranon Fractures in the Elderly
Brief Title: A Trial of Non-operative Versus Operative Management of Olecranon Fractures in the Elderly
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Complication rate in operative group on interim analysis and safety monitoring.
Sponsor: Andrew D Duckworth (Other)
Responsible Party: Sponsor-Investigator, Andrew D Duckworth, StR, Royal Infirmary of Edinburgh
Organization: Royal Infirmary of Edinburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/R/OST/05
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Olecranon Fractures in the Elderly

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-operative (Other): Patients in the non-operative arm will be managed conservatively using a sling, or an above elbow lightweight cast if problems with pain, for 10-14 days post injury. Patients will then be allowed to mobilise as able.
  Interventions: Other: Non-operative
- Operative (Other): Patients in this arm will be managed operatively for their olecranon fracture using either tension band wiring or plate fixation.
  Interventions: Other: Operative

INTERVENTIONS:
Other: Non-operative — Patients in the non-operative arm will be managed conservatively using a sling, or an above elbow lightweight cast if problems with pain, for 10-14 days post injury. Patients will then be allowed to mobilise as able.
  Arms: Non-operative
Other: Operative — For those patients in the operative group, tension band wire of plate fixation will be employed depending on the choice of their supervising consultant. Following surgery, the post-operative assessment and course will be as per normal protocol for patients who are not in this study. Patients in the operative group will be immobilised depending on fracture fixation during surgery and the decision will be made by the treating surgeon. Physiotherapy will be arranged when required.
  Arms: Operative

SUMMARY:
Proximal forearm fractures comprise approximately 5% of all fractures, with olecranon fractures accounting for almost 20% of thes fractures. There is limited conclusive evidence regarding the optimal treatment and outcome of these fractures within the elderly population with one case series in the literature describing 13 patients. Our trial includes all patients equal to or over the age of 75yrs presenting to the Edinburgh and Fife Orthopaedic Trauma Units with an isolated olecranon fracture. Patients who consent to enrol in the trial will be randomised to operative fixation using one of two treatment methods. Patients in the nonoperative group will be place in a sling for two weeks and then allowed to mobilise under supervised physiotherapy as per normal protocol. For those patients in the operative group, tension band wire of plate fixation will be employed depending on the choice of their supervising consultant. Patients will be evaluated over a one year period following their treatment.

DETAILED DESCRIPTION:
Patients with undisplaced olecranon fractures can be treated non-operatively. The aims of treatment in displaced olecranon fractures are the restoration of function and stability to the elbow joint4. The technique employed should allow preservation and reconstruction of the articular surface with minimal associated complications. Tension-band wiring (TBW) is the most recognised and commonly used fixation method, although plate fixation and intramedullary screw fixation are noted alternatives. Potential problems with the TBW technique are wound breakdown, infection, prominent metalwork, malunion and non-union. Furthermore, plate fixation is considered to be superior in distal/comminuted/oblique fractures and fracture-dislocations, with superior fracture reduction and fixation results, as well as a lower rate of re-operation.

The above described fixation techniques can be employed in elderly people, although difficulties associated with fixation in osteoporotic bone, wound breakdown and other complications is reported. In these patients, fracture excision with advancement of the triceps is a viable option if fixation is deemed inappropriate. However, there is limited evidence to suggest that non-operative treatment of displaced olecranon fractures in these elderly patients may provide adequate functional results. In a case series of 13 patients (mean age 81.8 years, >5 mm fracture displacement) treated non-operatively for a displaced olecranon fracture, outcome scores were excellent in 11 patients and poor in one.

Research Aim To determine if any difference exists in outcome (primary measure - DASH score) after one year between non-operative management AND operative treatment for olecranon fractures in patients 75yrs or older (≥75yrs).

Methodology This trial involves identifying patients over the age of 75yrs (≥75yrs) presenting to the Edinburgh Orthopaedic Trauma Unit and Fife Orthopaedic Trauma Unit with an isolated olecranon fracture. Patients who consent to enrol in the trial will be randomised to one of two recognised treatment techniques - non-operative management in a collar and cuff for two weeks OR operative management using tension band wire fixation or plate fixation. The trial will commence once ethical approval is granted by the Lothian Research Ethics Committee.

All statistical analysis was/will be performed by Dr Rob Elton. Prior to the study a power analysis determined the number of patients required in each trial. The primary outcome measure will be the DASH score, a continuous variable that follows a normal (Gaussian-shaped) distribution. This study is designed to determine a clinically relevant mean difference of 10 points between the two cohorts at one year after enrolment. A power analysis indicated that a total sample size of 50 (25 in each group) subjects will provide 80% statistical power to detect significant differences (0.05) in DASH scores, assuming an effect size of 0.8 (mean difference of 10 points, standard deviation of 12 points) using an unpaired t-test. To account for a possible loss to follow-up of up to 25%, we anticipate enrolling 35 subjects in each cohort for a total sample size of 70 subjects. A p value of < 0.05 was considered statistically significant.

All patients presenting to the units with a fracture of the olecranon that satisfy the inclusion criteria will be invited to participate in our study. Vulnerable populations will not be recruited.

A qualified member of the on-call team will introduce the study to the patient and initiate informed consent. If the patient agrees, a research fellow (Trauma and Orthopaedic StR3 level), not involved with the patient's care will review the study protocol in detail and address any questions the patient may have. If the patient is willing to participate, the research fellow will complete the informed consent with the patient. Patients will be given a copy of the consent form, and be informed that their participation is voluntary and that they can withdraw at any time during the study without detriment to their normal care in any way. Patients may take as long as they like to consider participation, provided that they still meet all the eligibility criteria documented above. Patients that are willing to participate in this study will get the same care of their fracture as patients that decide not to participate in the study.

On enrolment, a data collection form will be started with demographic and injury-related information collected. Patients will be randomised (performed by Dr Rob Elton using closed opaque envelopes) into one of the two groups (non-operative or operative). Patients in the non-operative group will be placed in a collar and cuff for two weeks and allowed to mobilise under supervised physiotherapy as per normal protocol. Patients in this group can be placed in cast (~60 degrees of flexion) if pain is too severe. For those patients in the operative group, tension band wire of plate fixation will be employed depending on the choice of their supervising consultant. Following surgery, the post-operative assessment and course will be as per normal protocol for patients who are not in this study. Patients in the operative group will be immobilised depending on fracture fixation during surgery and the decision will be made by the treating surgeon. Physiotherapy will be arranged when required

All follow-up assessment will take place during follow-up visits initially with the treating consultant surgeon's team and a dedicated member of the research team. Radiographs and other diagnostic studies will be obtained at the discretion of the treating surgeon and will not differ from routine clinical care.

Follow-up assessment will be collected over a one year period (2 weeks, 6 weeks, 3 months, 6 months and one year). Routine follow-up in our institution for patients who have sustained an olecranon fracture that is managed operatively involves outpatient clinic reviews with radiographs at 2 weeks, 6 weeks, three months and six months. Therefore, one additional visit at 1 year is required for this study with no additional radiographs. Radiographs will only be performed at one year on clinical indication.

At each visit physical examination, treatment, complications and re-operation (e.g. hardware removal), for each patient will be recorded. A member of the research team, blinded to the treatment method by sticking plaster over the entry position, will undertake functional testing and assessment.

By statistically analysing the outcome scores in the two groups, I aim to better determine the optimal management of this fracture in this age group. Using univariate analysis and multivariate regression analysis I will determine significant (p<0.05) predictors of outcome in relation to functional outcome score (DASH at one year).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥75 years
* Minimal, moderate or severe fragmentation of the olecranon
* Within two weeks of olecranon fracture

Exclusion Criteria:

* Patients unable to give informed consent
* Associated fractures to the coronoid, radial head and/or distal humerus
* Associated ligamentous injury, dislocation or subluxation
* Open fractures

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-10; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
DASH | One year
  Patient reported outcome measure specific to upper limb - DASH questionnaire at one year post injury/surgery.

SECONDARY OUTCOMES:
Mayo Elbow Performance Index (MEPI | One year
  Completion of the Mayo Elbow Performance Index (MEPI), a physician rate scale of function will completed for all patients15. The MEPI is a validated hundred-point system based upon pain (forty five points), range of motion (twenty points), stability (ten points) and daily function (twenty five points). Categorical ratings are assigned as follows: ninety to one hundred points is rated excellent; seventy-five to eighty-nine, good; sixty to seventy-four, fair; and less than sixty points, poor.
Range of motion | One year
  Range of motion at the elbow and forearm: will be measured using a standard full circle goniometer. Flexion, extension, supination and prontation will be measured in triplicate and the mean recorded to minimise intra-observer bias.
Pain | One year
  Pain assessment on an analogue scale 1-10.
Time taken to return to activities | One year
  Time taken to return to activities of daily living/work/sport
Radiographic Assessment | Six months
  Radiographic assessment used standard anteroposterior (AP) and lateral radiographs of the elbow. Outcome will also be assessed in detail with regards to loss of fracture reduction, complications, union and the development of radiographic degenerative changes +/- pseudoarthrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M McQueen, MD, FRCSEd, Principal Investigator — Edinburgh Orthopaedic Trauma Unit
Locations (2):
- United Kingdom (2):
  - Department of Orthopaedic Surgery, Fife (Dunfermline and Kirkcaldy), Dunfermline, Fife
  - Edinburgh Orthopaedic Trauma Unit, Edinburgh, Lothian

IPD SHARING:
Plan to Share IPD: Yes
Peer reviewed publication - undergoing review

REFERENCES:
- [Background] Rommens PM, Kuchle R, Schneider RU, Reuter M. Olecranon fractures in adults: factors influencing outcome. Injury. 2004 Nov;35(11):1149-57. doi: 10.1016/j.injury.2003.12.002. PMID 15488508
- [Background] Villanueva P, Osorio F, Commessatti M, Sanchez-Sotelo J. Tension-band wiring for olecranon fractures: analysis of risk factors for failure. J Shoulder Elbow Surg. 2006 May-Jun;15(3):351-6. doi: 10.1016/j.jse.2005.08.002. PMID 16679238
- [Background] Macko D, Szabo RM. Complications of tension-band wiring of olecranon fractures. J Bone Joint Surg Am. 1985 Dec;67(9):1396-401. PMID 3908460
- [Background] Horne JG, Tanzer TL. Olecranon fractures: a review of 100 cases. J Trauma. 1981 Jun;21(6):469-72. PMID 7230301
- [Background] Newman SD, Mauffrey C, Krikler S. Olecranon fractures. Injury. 2009 Jun;40(6):575-81. doi: 10.1016/j.injury.2008.12.013. Epub 2009 Apr 23. PMID 19394931
- [Background] Gartsman GM, Sculco TP, Otis JC. Operative treatment of olecranon fractures. Excision or open reduction with internal fixation. J Bone Joint Surg Am. 1981 Jun;63(5):718-21. PMID 7240294
- [Background] Parker MJ, Richmond PW, Andrew TA, Bewes PC. A review of displaced olecranon fractures treated conservatively. J R Coll Surg Edinb. 1990 Dec;35(6):392-4. PMID 2086804
- [Background] Veras Del Monte L, Sirera Vercher M, Busquets Net R, Castellanos Robles J, Carrera Calderer L, Mir Bullo X. Conservative treatment of displaced fractures of the olecranon in the elderly. Injury. 1999 Mar;30(2):105-10. doi: 10.1016/s0020-1383(98)00223-x. PMID 10476278